CLINICAL TRIAL: NCT06573320
Title: Investigating the Effect of Exercise on Clinical Symptoms, Cognitive Performance, and Quality of Life in Schizophrenia Patients Treated With Clozapine
Brief Title: Effect of Exercise on Clinical Symptoms, Cognitive Performance, and Quality of Life in Schizophrenia Patients Treated With Clozapine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Professor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Keah
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Clozapine; Exercise
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical exercise group (Experimental): physical exercise
  Interventions: Other: physical exercise
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: physical exercise — physical exercise
  Arms: physical exercise group

SUMMARY:
This prospective study aims to investigate the effects of exercise on clinical symptoms, cognitive performance, and quality of life in schizophrenia patients treated with Clozapine.

DETAILED DESCRIPTION:
The first developed atypical antipsychotic is clozapine. Its efficacy has been demonstrated in individuals with schizophrenia who have insufficient response to other antipsychotic therapies; nonetheless, its adverse effect profile is extensive. Among the antipsychotic medications now available, clozapine is not utilized as a first-line therapy because of major side effects such agranulocytosis. Increased salivation, sleepiness, weight gain, changes in blood pressure (sometimes an increase, sometimes a drop), elevated heart rate, dizziness, exhaustion, constipation, fever, and nocturnal enuresis are common adverse effects of clozapine usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated who were diagnosed with schizophrenia according to DSM-V criteria by psychiatrist at the Turkish Ministry of Health Kartal Dr. Lütfi Kırdar City Hospital
* using a therapeutic dose of 300-500 mg/day of clozapine,

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-08-26 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 12 weeks
  OCA is a short cognitive assessment method developed to detect particularly mild stages of cognitive impairment.
Positive and Negative Syndrome Scale (PANSS) | 12 weeks
  To evaluate clinical symptoms, both the exercise and control groups will be assessed by using the Positive and Negative Syndrome Scale (PANSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No